CLINICAL TRIAL: NCT05251688
Title: Effect of Cryoanalgesia on Reducing Unconscious Patients' Pain During Arterial Puncture
Brief Title: Cryoanalgesia for Arterial Puncture Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, sara Elsayed Ali Hegazy, Assistant Lecturer, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Cryoanalgesia
Record Dates: First submitted 2022-01-31; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Cryotherapy Effect

STUDY DESIGN:
Intervention Model Description: A quasi-experimental research design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Other): The participants were encountered two times (before and after the application of cryoanalgesia).
  Interventions: Other: Cryoanalgesia

INTERVENTIONS:
Other: Cryoanalgesia — On the first day of the study, the PI met the participants and assessed their level of consciousness using the Modified Glasgow Coma Scale to ensure that they were unconscious and reviewed the medical records to collect their sociodemographic data. After that, the participants received routine care before the arterial puncture. The PI assessed their pain scores during the puncture.
  In the second meeting (on the same day or the following day), the PI prepared the ice packs by crushing small pieces of ice and wrapping them in smooth gauze to avoid skin damage and moisture in the puncture area. Before the arterial puncture, the ice pack was applied over the selected puncture site (radial, brachial, or femoral artery) for 5 minutes in addition to the routine care. After removing the ice pack, the nurse palpated the artery, wiped of the residue of ice vapor present on the skin, and took the arterial blood sample. During the puncture, the PI assessed the participants' pain scores.

SUMMARY:
Arterial puncture is a painful procedure performed to assess patients' acid-base and respiratory status. Pain is a stressful situation for unconscious patients as they cannot communicate their feeling verbally. To control patients' pain and avoid the adverse effects of painkillers, nonpharmacological pain management strategies have been solicited. therefore, this study aimed to investigate the effect of cryoanalgesia on unconscious patients' pain during arterial puncture.

DETAILED DESCRIPTION:
Pain is a disturbing experience for patients in intensive care units (ICUs). It has deleterious effects on patients' health as it can lead to adverse physiological and psychological consequences. Patients undergo a wide variety of painful, invasive procedures to maintain their lives, such as arterial puncture, tracheal intubation, suctioning, insertion or removal of a chest tube, and wound care. A recent study recorded that the prevalence of pain in the ICU is approximately 31%. Another study reported that pain occurred in 5.0% -31.1% of the patients during the first 6 days of their stay in the ICU. Moreover, other studies have illustrated that the severity of pain increases significantly from the baseline during clinical procedures.

Arterial blood gases analysis is frequently requested for critically ill patients to diagnose and manage their acid-base imbalances and respiratory problems. Insertion of arterial lines for the purpose of repeated sampling is not practiced in many places for lack of monitoring devices or lack of expertise. Thus, arterial blood sampling is inevitable for these patients. Arterial samples can be obtained from different arteries such as the radial, brachial, femoral, axillary, dorsalis pedis, and posterior tibial. Regardless which site is used, all of these arteries have a high nerve supply and require deep needle insertion to access them. Hence, this procedure is usually associated with significant pain.

Managing procedural pain is a challenging task in ICUs as most patients have a reduced level of consciousness (LOC). Thus, they cannot express their pain and suffering, which can be disturbing situations for them that have adverse effects on their health. Therefore, when caring for unconscious patients, procedural pain must be evaluated and alleviated to avoid its physiological complications and prevent more intense pain.

In ICUs, pain management is mainly dependent on pharmacological and nonpharmacological interventions. Several pharmacological interventions are available, such as opioids, non-opioids, and adjunct analgesics. Although these medications are effective and fast, they have many adverse effects, including tolerance, suppression of cough reflexes, respiratory depression, immunosuppression, increased ICU stay, and worse post-ICU patient outcomes, especially for mechanically ventilated patients. Therefore, pharmacological interventions should not be the only option for pain management.

Nonpharmacological interventions are also advocated to minimize patients' pain because they are simple, safe, noninvasive, and inexpensive. They include relaxation techniques, cognitive-behavioral strategies, and biophysical interventions such as massage, pressure, and cutaneous electrical nerve stimulation by heat or cold application.

Cryoanalgesia is one of the most common nonpharmacological interventions. It is based on using low temperatures to produce analgesia or anesthesia. It slows the transmission of pain signals, increases the pain threshold, and provides anesthesia or numbness of the selected skin area. Fortunately, the nerve cells remain intact, allowing the nerves to regenerate and regain their normal function over time. Various cooling modalities can be used, such as ice packs, ice massage, cold water immersion, frozen gel packs, and vapocoolants.

Despite its benefits, prolonged repetitive ice application can lead to damage of the myelinated motor and sensory nerves. The myelin sheath is rich in lipids, and the ice results in the solidification and hardening of these lipids that may lead to the arrest of motor and sensory nerve conduction. It can also cause discomfort, frostbite, shivering, and changes in skin colour such as redness. So, it should be removed if the patient developed new pain, numbness, redness, or paleness of the application site. Cryoanalgesia should not be used for patients with severe hypoxia, traumatic brain injury, peripheral vessel disease, Raynaud's disease, diabetic neuropathy, and patients who are taking aspirin, anticoagulant, NSAID, and vasoactive agent. Additionally, it should be used in caution with people extreme age (infant, children, and elderly) as youngster have a thin layer of skin leading to skin breakdown and the elderly may become less sensitive to pain leading to burning. Moreover, open wound and stomas are among the situations that increase the risk of harm associated with using cold application as subcutaneous and deep tissues are more sensitive to temperature changes.

Cryoanalgesia is fast becoming a popular tool for controlling procedural pain as previous investigations have shown its benefits in decreasing pain during ICU procedures such as chest tube removal. Other researchers recorded its effectiveness in controlling pain associated with procedures involving the use of needles such as intramuscular injection, puncture of hemodialysis fistula, and immunization injection.

Additionally, several studies have investigated the effects of cryoanalgesia on pain during arterial puncture and reported its efficiency. However, empirical research on the effect of cryoanalgesia in reducing unconscious patients' pain remains scarce.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who were ≥18years old and were unconscious according to the Modified Glasgow Coma Scale (MGCS)

Exclusion Criteria:

* Sedated patients and those who were on controlled mode mechanical ventilation (MV). Patients who had traumatic brain injuries or Raynaud's syndrome were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
reducing pain intensity for unconscious patients during arterial puncture | pain intensity was assessed for two days
  Unconscious patients' pain was assessed during the arterial puncture before and after application of cryoanalgesia using the behavioral pain scale. This scale was adopted from Chanques et al. (2009). It was used to assess the participants' pain. The original behavioral pain scale was developed by Payen et al. (2001) to assess pain for intubated and mechanically ventilated patients. It consists of three items: facial expressions, movements of the upper limbs, and compliance with MV with a score range from 3 (no pain) to 12 (severe pain). Later on, Chanques et al. (2009) adapted the original BPS to facilitate pain assessment for non-intubated or non-ventilated patients who were unable to self-report their pain. They switched the "compliance with ventilation" domain of the initial BPS to a "vocalization" domain in this new form of BPS and combined it with the two other parts. The total score still ranges from 3 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hegazy, Principal Investigator — Faculty of Nursing, Mansoura University
Locations (1):
- Faculty of Nursing, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided